CLINICAL TRIAL: NCT07388706
Title: The Effect of Body Composition on Pain Threshold, Posture, Cervical Range of Motion, Sensation, and Cervical Function in Individuals With Non-Specific Neck Pain
Brief Title: Body Composition and Cervical Outcomes in Non-Specific Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Betül Taşpınar, Prof.Dr., Izmir Democracy University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Non-Specific Neck Pain-35
Record Dates: First submitted 2026-01-13; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Neck Pain
Keywords: Non-Specific Neck Pain; Body Composition; Cervical Range of Motion; Posture
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-Specific Neck Pain Group (Other): Participants diagnosed with non-specific neck pain
  Interventions: Other: Clinical Assessment

INTERVENTIONS:
Other: Clinical Assessment — Participants will undergo clinical assessments including body composition, pain threshold, posture, cervical range of motion, sensory function, and cervical disability. No therapeutic intervention will be applied.

SUMMARY:
Non-specific neck pain (NSNP) is a common musculoskeletal condition that significantly affects quality of life, daily activities, and work productivity. Although various physical, postural, and psychosocial factors have been associated with NSNP, the role of body composition in pain and functional outcomes remains unclear. Emerging evidence suggests that muscle and fat mass may influence musculoskeletal pain and related dysfunctions; however, studies examining these relationships in individuals with NSNP using objective measurements are limited. The purpose of this study is to investigate the effects of body composition on pain threshold, posture, cervical range of motion, sensation, and cervical function in individuals with non-specific neck pain. Individuals diagnosed with NSNP will be recruited from the Physical Medicine and Rehabilitation outpatient clinic. Participants' body composition, pain threshold, posture, cervical range of motion, sensory function, and cervical disability will be assessed using validated and objective measurement tools. Understanding the relationship between body composition and cervical outcomes in individuals with non-specific neck pain may contribute to early identification of risk factors and support the development of more targeted and effective physical therapy and rehabilitation strategies.

DETAILED DESCRIPTION:
Non-specific neck pain (NSNP) is defined as pain located in the posterior and lateral regions of the neck between the superior nuchal line and the first thoracic vertebra, in the absence of neurological or specific pathologies such as fracture, infection, or inflammation. Neck pain is a common and widespread condition with an episodic course that affects a large proportion of the population. It has been reported that at least 80% of individuals experience neck pain and related disorders at some point during their lifetime. Moreover, 30-50% of the general adult population report experiencing neck pain at least once per year. In addition, approximately 25% of outpatient visits to Physical Medicine and Rehabilitation clinics are due to neck pain complaints. For the majority of patients, neck pain is a complex biopsychosocial disorder accompanied by both physical and psychological symptoms. A relationship between the severity of neck pain and disability has been reported, and neck pain has been associated with decreased health-related quality of life, reduced work productivity, limitations in daily activities, and increased utilization of healthcare services. Risk factors for NSNP include prolonged and/or improper computer use, non-ergonomic desk and chair use, physical activity level, poor posture, body mass index (BMI), female sex, longer working hours, fewer hours of sleep, and stress. Body composition refers to the different tissues that make up total body mass, generally expressed as muscle, fat, bone, and residual mass. Analyses of muscle and fat tissues have shown that muscle cells consist of approximately 70% water, 7% fat, and 22% protein. An excess of fat cells in the body exerts an inhibitory effect on muscles, limiting their ability to function effectively and consequently restricting movement. Additionally, in physical fitness assessments, body composition is often evaluated by examining fat mass and fat-free mass. The literature reports that the load applied to the cervical spine is approximately 10-12 lbs when the head is in a neutral position, increasing to 60 lbs when the head is flexed to 60 degrees. Prolonged maintenance of a forward head position results in irritation of the facet joints, ligaments, and soft tissues of the cervical region. This irritation may cause neck pain radiating to the shoulders and upper back. Furthermore, sustained forward head posture may lead to trigger point formation in muscles, joint motion restrictions, disc degeneration, and potential pathologies such as cervical degenerative disc disease, cervical osteoarthritis, or cervical disc herniation. Maintaining proper posture has been identified as an important factor in the management of neck pain.

Chronic neck pain is a multifactorial condition associated not only with various dysfunctions in the cervical region but also with related structures in other parts of the body. In individuals with chronic neck pain, decreased muscle strength and endurance, limitations in joint range of motion, altered muscle activation patterns, forward head posture, impaired proprioception, and psychological dysfunctions have been reported. In chronic neck pain, a reduction in joint position sense and imbalance in the axio-scapular muscles lead to a shift in the body's midline. An anterior shift of the midline results in abnormal postural patterns, primarily forward head posture. This condition contributes to the development of upper crossed syndrome, which encompasses a range of postural impairments including shoulder elevation and protraction, upper thoracic kyphosis (dowager's hump), scapular winging, and reduced thoracic mobility.

Individuals with neck pain may present with movement restrictions, pain, decreased cervical and thoracic segmental mobility, myotomal muscle weakness, postural abnormalities, numbness or paresthesia, reduced muscle flexibility, increased muscle tension accompanied by a predisposition to myofascial trigger point formation, decreased proprioception, reduced endurance of neck muscles, and impaired coordination. Cervical range of motion supports head and neck movement by contributing to head stabilization during activities of daily living and allowing head orientation in various directions. The literature has demonstrated a reduction in cervical range of motion in individuals with chronic neck pain, and this limitation has been reported to be associated with neck pain severity and cervical functional status.

Therefore, elucidating the pathology of such pain and its associated factors in terms of frequency and impact on daily life is of great importance, and several studies have been conducted to date to investigate these aspects. Nevertheless, many factors related to the pathology and associated parameters of this type of pain remain unclear. Recently, the relationship between body composition-including muscle and fat mass-and various health problems has been reported, and increasing evidence has emerged regarding the role of body composition in different health conditions. For example, increased fat mass combined with age-related muscle loss has been associated with a higher risk of disability and mortality. On the other hand, some researchers have reported associations between body composition and musculoskeletal pain, demonstrating that greater fat mass and reduced muscle mass as body composition factors are related to musculoskeletal pain. In light of this information, studies investigating the effects of body composition in individuals with non-specific neck pain appear to be limited, particularly with respect to the inclusion of objective measurements.

ELIGIBILITY:
Inclusion Criteria:

* To be between 18-65 years old
* To be diagnosed with non-specific neck pain
* Not having had any surgery related to the cervical region

Exclusion Criteria:

* Having a neurological and psychiatric problem that may affect evaluation methods
* Pregnancy and pregnancy suspected
* To be an elite athlete
* Having a malignant disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-10-14 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Total Body Weight | Baseline
  Total body weight (kg) will be measured using the Tanita BC-700 (Tanita, Japan) body composition analyzer, which uses single-frequency bioelectrical impedance analysis (BIA) technology.
Body Mass Index (BMI) | Baseline
  Body mass index (BMI, kg/m²) will be calculated automatically by the Tanita BC-700 based on measured body weight and participant-reported height entered into the device prior to measurement.
Total Body Fat Percentage | Baseline
  Total body fat percentage (%) will be assessed using the Tanita BC-700 body composition analyzer based on bioelectrical impedance analysis.
Lower Extremity Fat Percentage | Baseline
  Lower extremity fat percentage (%) will be measured using the Tanita BC-700 body composition analyzer.
Total Body Muscle Percentage | Baseline
  Total body muscle percentage (%) will be assessed using the Tanita BC-700 body composition analyzer.
Lower Extremity Muscle Percentage | Baseline
  Lower extremity muscle percentage (%) will be measured using the Tanita BC-700 body composition analyzer.
Assessment of Pain Threshold | Baseline
  Pressure pain threshold (PPT) will be evaluated to determine participants' pain sensitivity. A Wagner digital algometer (Wagner Instruments) will be used for PPT assessment. Participants will be seated on a height-adjustable chair with their feet flat on the floor and knees flexed at 90 degrees. The algometer will be applied to the measurement sites at a 90-degree perpendicular angle. Measurements will be taken bilaterally at the following locations: lateral aspect of the C5 spinous process, the midpoint of the upper trapezius, and the midpoint of the deltoid muscle. Each site will be measured three times, with at least a 30-second interval between repeated measurements to prevent sensitization. The value at which the participant first perceives pain will be recorded, and the average of the three measurements will be calculated for each site.
Assessment of Posture | Baseline
  Posture will be evaluated using the New York Posture Rating Scale (NYPRS). This scale was first published in 1958 and assesses the body in 13 different regions for potential postural deviations. Each region is scored as follows: 5 points for correct posture, 3 points for moderate deviation, and 1 point for severe deviation. The total score ranges from 13 to 65 points, with higher scores indicating better overall posture.
Assessment of Cervical Range of Motion | Baseline
  Cervical range of motion (CROM) will be assessed using the Pa Crom Basic - Cervical Range of Motion device. The CROM device is an inclinometer system that relies on gravity and magnetic fields. It consists of two fixed inclinometers for the sagittal and frontal planes, a horizontal-plane inclinometer with a magnetic needle attached to the top of the device, an arm with a ruler for linear measurements, a magnetic cervical collar, and a vertebra-locating arm with a level system. The device is worn like a pair of glasses, resting on the nose, above both ears, and on the forehead. Flexion and extension movements are measured using the inclinometer positioned at the left lateral side of the head, right and left lateral flexion are measured with the inclinometer at the midpoint of the forehead, and right and left rotation movements are measured with the inclinometer on top of the head combined with the magnetic stabilizer.
Assessment of Sensation | Baseline
  Sensation will be assessed using the Semmes-Weinstein Monofilament Test, which evaluates light touch and pressure perception. The therapist applies monofilaments of increasing force (0.086-448 g) from the smallest detectable filament. Testing is performed on the first to fifth fingers, distal to proximal, on anterior and posterior surfaces. The pressure at which the patient first perceives the stimulus is recorded. Responses are marked on a hand map and classified using a color-coded system.
Assessment of Cervical Function | Baseline
  Cervical function will be evaluated using the Neck Disability Index (NDI). This questionnaire is used to assess pain originating from the neck and the degree of limitation in daily living activities. It was developed by Dr. Howard in 1980 and consists of a total of 10 items. These items cover areas such as pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleep, and recreation, with each item having six response options. Items are scored from 0 to 5, where 0 indicates no disability and 5 indicates complete disability. The total score can reach 50 points, which is then converted to a percentage. Higher scores indicate a higher level of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Sezgi KIZILIRMAK KARATAŞ, asst.prof., Principal Investigator — Izmir Democracy University; Onur Engin, asst.prof., Principal Investigator — Izmir Democracy University; Öykü Dündar, std., Principal Investigator — Izmir Democracy University; Büşra Aydın, Std., Principal Investigator — Izmir Democracy University; Turna Sümen, std., Principal Investigator — Izmir Democracy University; Nalan Anık, std., Principal Investigator — Izmir Democracy University; Kader İliman, std., Principal Investigator — Izmir Democracy University; Fadıma Kılıç, std., Principal Investigator — Izmir Democracy University
Locations (1):
- Betül TAŞPINAR, Konak, İ̇zmi̇r, Turkey (Türkiye)